CLINICAL TRIAL: NCT06468228
Title: A Phase 3 Multicenter, Randomized, Double-Blind Placebo-Controlled Study to Evaluate the Efficacy and Safety of Lutikizumab in Adult and Adolescent Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Assess Disease Activity and Safety of Lutikizumab in Adult and Adolescent Participants With Moderate to Severe Hidradenitis Suppurativa
Acronym: Intrepid
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M20-465; 2024-510730-40-00 (Other: EU CT)
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — lutikizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Period 1 (Experimental): Participants will be randomized to either Lutikizumab Dose B at baseline followed by Lutikizumab Dose A, or a matching placebo dose equivalent for both, every week through Week 16 .
  Interventions: Drug: Lutikizumab; Drug: Placebo
- Period 2: Lutikizumab Every Week (Experimental): Participants randomized to lutikizumab in Period 1 who complete Week 16 of the study will be re-randomized to lutikizumab Dose A through Week 52
  Interventions: Drug: Lutikizumab
- Period 2: Lutikizumab Every Other Week (Experimental): Participants randomized to lutikizumab in Period 1 who complete Week 16 of the study will be re-randomized to lutikizumab Dose A every other week though week 52
  Interventions: Drug: Lutikizumab; Drug: Placebo
- Period 2: Placebo to Lutikizumab Group (Experimental): Participants randomized to Placebo in Period 1 who complete Week 16 of the study will initiate lutikizumab with Dose B followed by Dose A every week.
  Interventions: Drug: Lutikizumab
- Period 2: Placebo to Lutikizumab Group Every Week (Experimental): Participants that were assigned Placebo in Period 1 and initiated lutikizumab in Period 2 will then be re-randomized to lutikizumab Dose A every week through Week 52
  Interventions: Drug: Lutikizumab
- Period 2: Placebo to Lutikizumab Group Every Other Week (Experimental): The participants that were assigned Placebo in Period 1 and initiated lutikizumab in Period 2 will then be re-randomized to lutikizumab Dose A every other week through Week 52
  Interventions: Drug: Lutikizumab; Drug: Placebo
- Period 3: Open-label Lutikizumab (Experimental): Starting at Week 68 in Period 3, all participants will receive Open-label Lutikizumab every other week
  Interventions: Drug: Lutikizumab
- Sub-Study: Lutikizumab Pre-Filled Pen (Experimental): Lutikizumab solution for injection in prefilled pen (EOW) for 60 weeks, followed by lutikizumab solution for injection in prefilled syringes (EOW) for 96 weeks.
  Interventions: Drug: Lutikizumab

INTERVENTIONS:
Drug: Lutikizumab — Subcutaneous injection
  Other Names: ABT-981
Drug: Placebo — Subcutaneous injection
  Arms: Period 1; Period 2: Lutikizumab Every Other Week; Period 2: Placebo to Lutikizumab Group Every Other Week

SUMMARY:
Hidradenitis suppurativa (HS) is a chronic and often painful inflammatory skin disease which includes the forming of lumps, abscesses and scars in areas of the skin such as under the breasts, under armpits, inner thighs, groin and buttocks. This study will compare lutikizumab versus placebo for the treatment of adult and adolescent participants with the signs and symptoms of moderate to severe HS .

Lutikizumab is an investigational drug being developed for the treatment of HS. During Period 1 of the study, participants will placed in 1 of 2 groups called treatment arms. There is a 1 in 2 chance that participants will be assigned to placebo. Around 1280 adult and adolescent participants with moderate to severe HS will be enrolled in the study at approximately 275 sites world wide. During Period 2, participants that were part of the lutikizumab treatment arm in Period 1 will be re-randomized to 1 of 2 lutikizumab treatment arms. Participants that were part of the Placebo arm in Period 1 will start Period 2 with an initiation of lutikizumab followed by a re-randomization to 1 of 2 lutikizumab treatment arms.

In Period 1, participants will receive subcutaneous injections of lutikizumab or placebo every week for 16 weeks. In Period 2, participants that were randomized to lutikizumab in Period 1 will receive subcutaneous injections of lutikizumab every week or every other week for 36-weeks. Participants that were randomized to the placebo arm in Period 1 will receive subcutaneous injections of lutikizumab every week for 16 weeks, then either every week or every other week for 20 weeks.

Period 3 is the Long Term Extentsion (LTE) and through Week 68, participants will continue to receive lutikizumab SC using the same assigned dosing regimen from the end of Period 2 for 16 weeks followed by open-label lutikizumab EOW for 140 weeks.

Participants in the US that complete Periods 1 & 2 will have the option to enroll in a 156-week open-label Sub-Study that will assess the long term safety and efficacy of lutikizumab in a prefilled pen.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires and diaries.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe HS for at least 6 months prior to Baseline as determined by the investigator (i.e., through medical history and interview of participant).
* Total abscess and inflammatory nodule (AN) count of ≥ 5 at Baseline
* Hidradenitis suppurativa (HS) lesions present in at least two distinct anatomic areas at Baseline.
* At least 1 anatomic area of HS involvement characterized as Hurley Stage II or higher at Baseline.

Exclusion Criteria:

* Any evidence of Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Confirmed positive anti-HIV antibody (HIV Ab) test.
* Evidence of active tuberculosis or meets tuberculosis exclusionary parameter

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1280 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Hidradenitis Suppurative Clinical Response (HiSCR) 75 | At Week 16
  HiSCR 75 is defined as at least a 75% reduction from baseline in the total abscess and inflammatory nodule (AN) count, with no increase in abscess count and no increase in draining fistula count relative to baseline.
Number of Participants with Adverse Events (AEs) | Up to Approximately Week 62
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Numeric Rating Scale (NRS) 30 among Participants with Baseline NRS >=3 | At Week 8
  NRS 30 is defined as at least a 30% reduction and at least 1-unit reduction from Baseline in worst skin pain (maximal daily pain), as assessed by the Patient's Global Assessment (PGA) of Skin Pain.
Change from Baseline in Dermatology Life Quality Index (DLQI) among participants ≥ 16 years of age at Baseline | At Week 16
  DLQI (Dermatology Life Quality Index) assesses symptoms and impacts of dermatologic diseases on quality of life. DLQI scores range from 0 (no effect) to 30 (very large effect), with a higher score indicating a more impaired quality of life.
Change from Baseline in Hidradenitis Suppurativa Impact Assessment (HSIA) | At Week 16
  The HSIA is an 18-item PRO questionnaire developed to assess the impact of HS on the daily lives of subjects in the 7 days prior to the assessment. Items 1 - 16 of the HSIA are scored on a 0 to 10 NRS, where 0 represents no impact and 10 represents extreme impact.
Change from Baseline in Hidradenitis Suppurativa Symptom Assessment (HSSA) Worst Drainage Score | At Week 16
  The HSSA (24-hour recall) is a 9-item PRO questionnaire developed to assess the primary symptoms of Hidradenitis Suppurativa (HS) in the 7 consecutive days prior to assessments. Each item of the HSSA is scored on an 11-point (0 to 10) NRS, where 0 represents no symptoms and 10 represents extreme symptom experience.
Change from Baseline in number of Draining Fistulas Count among participants with at least 1 draining fistula at Baseline | At Week 16
Percentage of Participants Achieving HiSCR 90 | At Week 16
  HiSCR 90 is defined as at least a 90% reduction from baseline in the total abscess and inflammatory nodule (AN) count, with no increase in abscess count and no increase in draining fistula count relative to baseline.
Change from Baseline in the Patient's Global Assessment of HS-related Skin Pain (NRS) | At Week 8
Change from Baseline in HSSA | At Week 16
  The HSSA (24-hour recall) is a 9-item PRO questionnaire developed to assess the primary symptoms of Hidradenitis Suppurativa (HS) in the 7 consecutive days prior to assessments. Each item of the HSSA is scored on an 11-point (0 to 10) NRS, where 0 represents no symptoms and 10 represents extreme symptom experience.
Change from Baseline in the Patient's Global Assessment of HS-related Odor (smell), based on the HSSA Question 8 | At Week 16
  The HSSA (24-hour recall) is a 9-item PRO questionnaire developed to assess the primary symptoms of HS in the 7 consecutive days prior to assessments. Each item of the HSSA is scored on an 11-point (0 to 10) NRS, where 0 represents no symptoms and 10 represents extreme symptom experience.
Percentage of Participants with an Occurrence of HS Flare in Period 1 | Baseline to Week 16
  HS Flare is defined as at least one occurrence of a ≥ 25% increase in AN count with a minimum absolute increase of 2 relative to Baseline.
Change from Baseline in Hidradenitis Suppurativa Impact Assessment (HSIA) Emotional Domain | At Week 16
Change from Baseline in HSIA Mobility Domain | at Week 16

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (274):
- United States (72):
  - Cahaba Dermatology & Skin Health Center /ID# 263795, Birmingham, Alabama
  - Medical Dermatology Specialists /ID# 263394, Phoenix, Arizona
  - Banner University Medicine Dermatology /ID# 263557, Tucson, Arizona
  - Dermatology Trial Associates /ID# 264587, Bryant, Arkansas
  - Arkansas Research Trials /ID# 263901, North Little Rock, Arkansas
  - Private Practice - Dr. Tooraj Raoof /ID# 263756, Encino, California
  - NorCal Medical Research /ID# 279008, Greenbrae, California
  - Dermatology Research Associates - Los Angeles /ID# 263765, Los Angeles, California
  - Stanford University School of Medicine - Redwood City /ID# 263711, Redwood City, California
  - Integrative Skin Science and Research /ID# 264600, Sacramento, California
  - Clinical Trials Research Institute /ID# 263743, Thousand Oaks, California
  - Clearlyderm Dermatology - West Boca /ID# 265023, Boca Raton, Florida
  - Apex Clinical Trials /ID# 263815, Brandon, Florida
  - TrueBlue Clinical Research /ID# 265041, Brandon, Florida
  - Florida Academic Dermatology Center /ID# 263834, Coral Gables, Florida
  - Direct Helpers Research Center /ID# 278343, Hialeah, Florida
  - Skin Care Research - Hollywood /ID# 263805, Hollywood, Florida
  - GSI Clinical Research, LLC /ID# 263827, Margate, Florida
  - Sullivan Dermatology /ID# 263511, Miami, Florida
  - Vitalia Medical Research /ID# 278321, North Palm Beach, Florida
  - Renstar Medical Research - Ocala - Northeast 1st Avenue /ID# 263842, Ocala, Florida
  - Skin Care Research - Tampa /ID# 263819, Tampa, Florida
  - Advanced Clinical Research Institute /ID# 263808, Tampa, Florida
  - University of South Florida /ID# 269624, Tampa, Florida
  - Alliance Clinical Research of Tampa /ID# 264594, Tampa, Florida
  - TruDerm Research /ID# 278217, Wellington, Florida
  - Centricity Research Columbus Dermatology /ID# 266530, Columbus, Georgia
  - Cleaver Medical Group Dermatology /ID# 263845, Dawsonville, Georgia
  - Treasure Valley Medical Research /ID# 263671, Boise, Idaho
  - DeNova Research /ID# 264593, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine /ID# 265007, Chicago, Illinois
  - Arlington Dermatology /ID# 263410, Rolling Meadows, Illinois
  - Dawes Fretzin, LLC /ID# 264601, Indianapolis, Indiana
  - Dermatology Partners of Leawood /ID# 263533, Leawood, Kansas
  - Equity Medical, LLC /ID# 268590, Bowling Green, Kentucky
  - Dermatology Specialists Research (DS Research) - Kentucky /ID# 263343, Louisville, Kentucky
  - Tulane University School of Medicine /ID# 263899, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center /ID# 263709, Boston, Massachusetts
  - UMass Memorial Medical Center /ID# 274149, Worcester, Massachusetts
  - Hamzavi Dermatology - Canton /ID# 263538, Canton, Michigan
  - Michigan Center for Medical Research /ID# 263547, Clarkston, Michigan
  - Michigan Center for Skin Care Research /ID# 267228, Clinton Township, Michigan
  - Dermatology and Skin Center of Lees Summit /ID# 263567, Lee's Summit, Missouri
  - MediSearch Clinical Trials /ID# 263582, Saint Joseph, Missouri
  - Vivida Dermatology- Flamingo /ID# 263716, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center - Old Etna Road /ID# 263713, Lebanon, New Hampshire
  - StracSkin, PLLC /ID# 263387, Portsmouth, New Hampshire
  - Mount Sinai Doctors - Dermatology /ID# 264602, New York, New York
  - Wake Forest University Baptist Medical Center (WFUBMC) /ID# 264507, Winston-Salem, North Carolina
  - Dermatology of Greater Columbus /ID# 263497, Bexley, Ohio
  - University Hospitals Cleveland Medical Center /ID# 263600, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center - CarePoint East /ID# 263598, Columbus, Ohio
  - Dermatologists of Southwest Ohio - Mason /ID# 263588, Mason, Ohio
  - Apex Clinical Research Center /ID# 272787, Mayfield Heights, Ohio
  - Dermatology Partners /ID# 264999, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center /ID# 264590, Pittsburgh, Pennsylvania
  - Clinical Research Center of the Carolinas /ID# 263407, Charleston, South Carolina
  - Medical University of South Carolina /ID# 263890, Charleston, South Carolina
  - ADCS - Spartanburg /ID# 267207, Spartanburg, South Carolina
  - Arlington Research Center, Inc /ID# 263895, Arlington, Texas
  - Bellaire Dermatology Associates /ID# 263850, Bellaire, Texas
  - Studies in Dermatology LLC /ID# 263399, Cypress, Texas
  - Reveal Research Institute - Dallas /ID# 267233, Dallas, Texas
  - Center for Clinical Studies - Houston - Binz Street /ID# 263378, Houston, Texas
  - Texas Dermatology Research Center /ID# 264488, Plano, Texas
  - Texas Dermatology and Laser Specialists /ID# 263778, San Antonio, Texas
  - The Woodlands Dermatology Associates /ID# 266820, The Woodlands, Texas
  - Dermatology Associates of Tyler /ID# 265002, Tyler, Texas
  - University of Utah /ID# 263818, Murray, Utah
  - Virginia Clinical Research /ID# 264553, Norfolk, Virginia
  - Frontier Dermatology /ID# 278387, Mill Creek, Washington
  - Dermatology Specialists of Spokane /ID# 264499, Spokane, Washington
- Argentina (4):
  - Consultorios Reumatologicos Pampa /ID# 265911, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto De Investigaciones Clínicas Córdoba /ID# 264297, Córdoba, Córdoba Province
  - Instituto de Especialidades de la Salud Rosario - Clinica del Torax /ID# 266132, Rosario, Santa Fe Province
  - Buenos Aires Skin /ID# 264299, Buenos Aires
- Australia (5):
  - Paratus Clinical Research Woden /ID# 263125, Phillip, Australian Capital Territory
  - Momentum Clinical Research /ID# 263192, Darlinghurst, New South Wales
  - Premier Dermatology /ID# 263124, Kogarah, New South Wales
  - Veracity Clinical Research /ID# 263126, Woolloongabba, Queensland
  - Sinclair Dermatology - Melbourne /ID# 263121, East Melbourne, Victoria
- Austria (2):
  - Medizinische Universitaet Graz /ID# 263306, Graz, Styria
  - Medizinische Universitaet Wien /ID# 264043, Vienna
- Belgium (7):
  - Universite Libre de Bruxelles - Hopital Erasme /ID# 263097, Anderlecht, Brussels Capital
  - Cliniques Universitaires UCL Saint-Luc /ID# 263096, Brussels, Brussels Capital
  - Universitair Ziekenhuis Brussel /ID# 263101, Jette, Brussels Capital
  - Grand Hôpital de Charleroi - Les Viviers /ID# 263100, Charleroi, Hainaut
  - UZ Gent /ID# 263099, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 263098, Leuven, Vlaams-Brabant
  - CHU de Liege /ID# 263095, Liège
- Bosnia and Herzegovina (4):
  - Clinical Center University of Sarajevo - Bolnicka /ID# 265908, Sarajevo, Federation of Bosnia and Herzegovina
  - University Clinical Center Tuzla /ID# 265906, Tuzla, Federation of Bosnia and Herzegovina
  - Klinicki centar Banja Luka /ID# 265905, Banja Luka, Republika Srpska
  - Klinicki centar Banja Luka /ID# 265909, Banja Luka, Republika Srpska
- Bulgaria (6):
  - Acibadem City Clinic Tokuda Hospital /ID# 263300, Sofiya, Sofia
  - Ambulatory for Specialized Medical Care-IPSMC-skin and venereal diseases /ID# 262891, Sofiya, Sofia
  - Diagnostic Consultative Centre (Dcc) - Foкus 5 /ID# 262893, Sofiya, Sofia
  - Medical Center Hera EOOD /ID# 263010, Sofiya, Sofia
  - Medical Center Cordis /ID# 262894, Pleven
  - UMHAT Professor Stoyan Kirkovich /ID# 262892, Stara Zagora
- Canada (17):
  - Beacon Dermatology Inc /ID# 264262, Calgary, Alberta
  - Rejuvenation Dermatology - Edmonton Downtown /ID# 265963, Edmonton, Alberta
  - Stratica Dermatology /ID# 265856, Edmonton, Alberta
  - Interior Dermatology Centre - Probity - PPDS /ID# 266202, Kelowna, British Columbia
  - Brunswick Dermatology Center /ID# 264260, Fredericton, New Brunswick
  - Karma Clinical Trials /ID# 265962, St. John's, Newfoundland and Labrador
  - Skin Health /ID# 267735, Cobourg, Ontario
  - Leader Research /ID# 266114, Hamilton, Ontario
  - DermEffects /ID# 265262, London, Ontario
  - Derm Care Clinic /ID# 265261, Mississauga, Ontario
  - York Dermatology Clinic & Research Centre /ID# 265265, Richmond Hill, Ontario
  - FACET Dermatology /ID# 265267, Toronto, Ontario
  - Private Practice - Dr. Kim Papp Clinical Research /ID# 265266, Waterloo, Ontario
  - Centre de Recherche Saint-Louis /ID# 265855, Québec, Quebec
  - Private Practice - Dr. Angelique Gagne-Henley /ID# 264263, Saint-Jérôme, Quebec
  - SkinSense Dermatology /ID# 265964, Saskatoon, Saskatchewan
  - Diex Recherche Quebec Inc. /ID# 265263, Québec
- Chile (3):
  - Centro Internacional de Estudios Clinicos - CIEC /ID# 266129, Santiago, Region Metropolitana Santiago
  - Clinica Dermacross /ID# 266127, Vitacura, Region Metropolitana Santiago
  - Fundacion Innovacion Cardiovascular /ID# 264844, Independencia, Santiago Metropolitan
- Colombia (3):
  - Centro de Inmunología y Genética CIGE SAS /ID# 263793, Medellín, Antioquia
  - Centro de Investigacion en Reumatologia y especialidades Medicas S.A.S- CIREEM /ID# 265093, Bogotá, Cundinamarca
  - Healthy Medical Center S.A.S /ID# 265091, Zipaquirá, Cundinamarca
- Croatia (4):
  - Klinicki Bolnicki Centar Zagreb /ID# 263989, Grad Zagreb, City of Zagreb
  - Klinicki Bolnicki Centar Sestre Milosrdnice /ID# 265069, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Osijek /ID# 265916, Osijek, County of Osijek-Baranja
  - Specialty Hospital Medico /ID# 263922, Rijeka, Primorje-Gorski Kotar County
- Czechia (3):
  - Fakultni nemocnice Ostrava /ID# 264041, Ostrava, Ostrava-mesto
  - Karlovarska Krajska Nemocnice - Karlovy Vary /ID# 265354, Karlovy Vary
  - Fakultni nemocnice Kralovske Vinohrady /ID# 264040, Prague
- Denmark (3):
  - Herlev and Gentofte Hospital /ID# 265839, Hellerup, Capital Region
  - Aarhus Universitetshospital - Skejby /ID# 265657, Aarhus, Central Jutland
  - Roskilde Sygehus /ID# 274895, Roskilde, Region Sjælland
- France (6):
  - Hopital Edouard Herriot /ID# 263456, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire de Saint Etienne - Hopital Nord /ID# 263459, St-Priest-en-Jarez, Pays de la Loire Region
  - Cabinet medical - Le bateau Blanc /ID# 263465, Martigues, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Universitaire de Rouen (CHU)- Hopital Charles Nicolle /ID# 263995, Rouen, Seine-Maritime
  - Groupe Hospitalier Paris Saint-Joseph /ID# 263996, Paris
  - Polyclinique Courlancy /ID# 263313, Reims
- Germany (13):
  - Universitaetsklinikum Freiburg /ID# 263659, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen /ID# 271718, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 263075, Erlangen, Bavaria
  - Beldio Research GmbH /ID# 263074, Memmingen, Bavaria
  - Rosenpark Research /ID# 269202, Darmstadt, Hesse
  - Fachklinik Bad Bentheim /ID# 263067, Bad Bentheim, Lower Saxony
  - Universitaetsmedizin Rostock /ID# 278301, Rostock, Mecklenburg-Vorpommern
  - Katholisches Klinikum Bochum /ID# 262976, Bochum, North Rhine-Westphalia
  - Universitaetsklinikum Muenster /ID# 263068, Münster, North Rhine-Westphalia
  - Hautarztpraxis Mortazawi /ID# 271673, Remscheid, North Rhine-Westphalia
  - Hautarztpraxis Dr. Kirschner /ID# 263656, Mainz, Rhineland-Palatinate
  - HMS GmbH Zimmer /ID# 278634, Merzig, Saarland
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 263076, Berlin
- Greece (4):
  - University General Hospital Attikon /ID# 263413, Athens, Attica
  - General Hospital Andreas Syggros /ID# 263417, Athens, Attica
  - Hospital of Skin and Venereal Diseases- Thessaloniki /ID# 263416, Thessaloniki
  - Papageorgiou General Hospital /ID# 263415, Thessaloniki
- Guatemala (2):
  - Dermos S.A. /ID# 265857, Guatemala City
  - Prosalud /Id# 266586, Guatemala City
- Hungary (4):
  - Pécsi Tudományegyetem /ID# 264120, Pécs, Baranya
  - Debreceni Egyetem-Klinikai Kozpont /ID# 263423, Debrecen, Hajdú-Bihar
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz /ID# 263424, Kaposvár, Somogy County
  - Semmelweis Egyetem /ID# 263451, Budapest
- Ireland (4):
  - Our Lady of Lourdes Hospital - Drogheda /ID# 265893, Drogheda, Louth
  - South Infirmary Victoria University Hospital /ID# 265872, Cork
  - University College Dublin /ID# 265875, Dublin
  - Mater Misericordiae University Hospital /ID# 265914, Dublin
- Israel (7):
  - Rabin Medical Center /ID# 262992, Petah Tikva, Central District
  - HaEmek Medical Center /ID# 267297, Afula, Haifa District
  - Galilee Medical Center /ID# 262995, Nahariya, Northern District
  - The Chaim Sheba Medical Center /ID# 262993, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 266581, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus- Haifa /ID# 262994, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 262884, Jerusalem
- Italy (7):
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale S.Anna /ID# 263474, Cona, Ferrara
  - AZIENDA USL TOSCANA CENTRO - Ospedale Piero Palagi /ID# 263454, Florence, Firenze
  - IRCCS Istituto Clinico Humanitas /ID# 263503, Rozzano, Lombardy
  - Azienda Ospedaliera Universitaria Federico II /ID# 263539, Naples, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita Cattolica /ID# 263473, Rome, Roma
  - AOU Policlinico G. Rodolico - San Marco /ID# 263469, Catania
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 263471, Milan
- Japan (12):
  - Nagoya City University Hospital /ID# 263874, Nagoya, Aichi-ken
  - Fujita Health University Hospital /ID# 265440, Toyoake, Aichi-ken
  - Takagi Dermatological Clinic /ID# 264810, Obihiro-Shi, Hokkaido
  - Iwate Medical University Uchimaru Medical Center /ID# 273799, Morioka, Iwate
  - University Hospital Kyoto Prefectural University of Medicine /ID# 264291, Kyoto, Kyoto
  - Niigata University Medical & Dental Hospital /ID# 276568, Niigata, Niigata
  - University of the Ryukyus Hospital /ID# 264605, Ginowan-shi, Okinawa
  - Osaka Metropolitan University Hospital /ID# 265682, Osaka, Osaka
  - Kindai University Hospital /ID# 264322, Sakai-shi, Osaka
  - Dokkyo Medical University Saitama Medical Center /ID# 265400, Koshigaya, Saitama
  - Fukuoka University Hospital /ID# 263991, Fukuoka
  - Nihon University Itabashi Hospital /ID# 264661, Tokyo
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 277709, Kaunas
  - Vilnius University Hospital Santaros Klinikos /ID# 277707, Vilnius
- Mexico (4):
  - Grupo Clinico CATEI S C /ID# 265276, Guadalajara, Jalisco
  - Cryptex Investigación Clínica /ID# 265271, Mexico City, Mexico City
  - Eukarya PharmaSite /ID# 265307, Monterrey, Nuevo León
  - Sociedad de Metabolismo y Corazon S.C. /ID# 265915, Veracruz
- Erasmus Medisch Centrum /ID# 263377, Rotterdam, South Holland, Netherlands
- New Zealand (2):
  - Greenlane Clinical Centre /ID# 263191, Epsom, Auckland
  - Clinical Trials New Zealand /ID# 265432, Hamilton, Waikato Region
- Norway (3):
  - Stavanger Universitetssykehus /ID# 265997, Stavanger, Rogaland
  - Universitetssykehuset I Nord-Norge /ID# 265992, Tromsø, Troms
  - Oslo University Hospital - Rikshospitalet /ID# 265996, Oslo
- Poland (8):
  - Oftalmika sp. z o.o. /ID# 263087, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczny gabinet dermatologiczny Aplikacyjno-Badawczy Marek Brzewski, Paw /ID# 277221, Krakow, Lesser Poland Voivodeship
  - Centrum Nowoczesnych Terapii Dobry Lekarz sp.z.o.o. /ID# 263146, Krakow, Lesser Poland Voivodeship
  - Panstwowy Instytut Medyczny Mswia /Id# 277307, Warsaw, Masovian Voivodeship
  - Klinika Ambroziak Dermatologia /ID# 263173, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Angelius Provita /ID# 277204, Katowice, Silesian Voivodeship
  - DERMED Centrum Medyczne Sp. z o.o /ID# 263147, Lodz, Łódź Voivodeship
  - Santa Sp. z o..o. Santa Familia PTG Lodz /ID# 263181, Lodz, Łódź Voivodeship
- Portugal (4):
  - Unidade Local de Saude do Alto Ave, EPE /ID# 265158, Guimarães, Braga District
  - CUF Descobertas Hospital /ID# 263188, Lisbon, Lisbon District
  - Unidade Local de Saude de Sao Jose, EPE /ID# 265155, Lisbon
  - Unidade Local de Saude de Santo Antonio, E.P.E. /ID# 265479, Porto
- Puerto Rico (2):
  - Private Practice - Dr. Alma Cruz /ID# 263204, Carolina
  - Clinical Research Puerto Rico /ID# 263450, San Juan
- Romania (3):
  - Spitalul Clinic Colentina /ID# 263303, Bucharest, București
  - Private Practice - Dr. Orasan Remus /ID# 263305, Cluj-Napoca, Cluj
  - Centrul Medical Euromed /ID# 263304, Bucharest
- Saudi Arabia (2):
  - King Abdulaziz Medical City /ID# 266121, Jeddah, Mecca Region
  - King Saud University Med City /ID# 266120, Riyadh
- Serbia (4):
  - Military Medical Academy /ID# 263257, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 263256, Belgrade, Beograd
  - University Clinical Center Kragujevac /ID# 264211, Kragujevac, Sumadijski Okrug
  - University Clinical Center Vojvodina /ID# 263260, Novi Sad
- Singapore (2):
  - National University Hospital /ID# 264673, Singapore
  - National Skin Centre /ID# 264680, Singapore
- Slovakia (4):
  - Poliklinika Bezrucova (Cliniq s.r.o.) /ID# 263921, Bratislava, Bratislava Region
  - Univerzitna nemocnica L. Pasteura Kosice /ID# 263907, Košice, Košice Region
  - Fakultna nemocnica s poliklinikou Nove Zamky /ID# 265944, Nové Zámky, Nitra Region
  - Fakultna nemocnica Trnava /ID# 263905, Trnava
- Slovenia (2):
  - University Medical Centre Ljubljana /ID# 265720, Ljubljana
  - University Medical Centre Maribor /ID# 265827, Maribor
- South Africa (4):
  - Global Clinical Trials /ID# 262839, Pretoria, Gauteng
  - Life Chatsmed Garden Hospital /ID# 270237, Chatsworth, KwaZulu-Natal
  - Ahmed Al-Kadi Private Hospital /ID# 262837, Durban, KwaZulu-Natal
  - Dr Ahmed Ismail Manjra /ID# 262838, Westville, KwaZulu-Natal
- South Korea (9):
  - Pusan National University Hospital /ID# 271496, Busan, Busan Gwang Yeogsi
  - SoonChunHyang University Hospital Cheonan /ID# 271320, Cheonan-si, Chungcheongnam-do
  - Korea University Ansan Hospital /ID# 264227, Ansan-si, Gyeonggido
  - CHA Bundang Medical Center /ID# 264225, Seongnam, Gyeonggido
  - Yonsei University Health System Severance Hospital /ID# 271353, Seoul, Seoul Teugbyeolsi
  - SoonChunHyang University Seoul Hospital /ID# 264224, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 264228, Seoul, Seoul Teugbyeolsi
  - Hallym University Kangnam Sacred Heart Hospital /ID# 264226, Seoul, Seoul Teugbyeolsi
  - The Catholic University Of Korea, Eunpyeong St. Mary'S Hospital /ID# 271348, Seoul
- Spain (6):
  - Hospital Universitari Parc Tauli /ID# 262942, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla /ID# 263039, Santander, Cantabria
  - Hospital Universitario Virgen de la Victoria /ID# 262941, Málaga, Malaga
  - Hospital de Manises /ID# 262938, Manises, Valencia
  - Hospital General Universitario Gregorio Maranon /ID# 262940, Madrid
  - Consorci Hospital General Universitario de Valencia /ID# 262944, Valencia
- Sweden (2):
  - Karolinska University Hospital Solna /ID# 264530, Solna, Stockholm County
  - Universitetssjukhuset Örebro /ID# 265064, Örebro, Örebro County
- Switzerland (4):
  - University Hospital Basel /ID# 264245, Basel Town, Canton of Basel-City
  - Dermatology & Skin Care Clinic /ID# 264030, Buochs, Canton of Nidwalden
  - Kantonsspital St.Gallen /ID# 264238, Sankt Gallen, Canton of St. Gallen
  - University Hospital Zurich /ID# 266142, Zurich, Canton of Zurich
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 264619, Kaohsiung City, Kaohsiung
  - Taichung Veterans General Hospital /ID# 270741, Taichung
  - National Taiwan University Hospital /ID# 264618, Taipei
  - Mackay Memorial Hospital /ID# 263661, Taipei
  - Taipei Veterans General Hospital /ID# 265879, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 264620, Taoyuan
- United Kingdom (8):
  - Royal Cornwall Hospital /ID# 277507, Truro, Cornwall
  - Queen Margaret Hospital /ID# 264198, Dunfermline, Fife
  - Gloucestershire Royal Hospital /ID# 265848, Gloucester, Gloucestershire
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 264121, London, Greater London
  - Harrogate District Hospital /ID# 265632, Harrogate, North Yorkshire
  - Southlands Hospital /ID# 276976, Shoreham-by-Sea, West Sussex
  - Bristol Royal Infirmary /ID# 263937, Bristol
  - Royal Victoria Infirmary /ID# 273368, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M20-465